CLINICAL TRIAL: NCT05617391
Title: An Evaluation of Concordance of Smartwatch ECG and One Clinical ECG and Comparison of The Two ECGS in Terms of Predictive Risks
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WATCH4ECG
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Childhood Cancer; Cardiomyopathy, Primary
MeSH Terms: conditions — Neoplasms; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Childhood Cancer Survivors: The comparison of two ECGs in terms of predictive risk.

SUMMARY:
The participant is being asked to take part in this trial, because the participant is a survivor of childhood cancer.

Primary Objective

To evaluate remote cardiomyopathy prediction via smartwatch and one clinical ECG and assess the concordance of the two ECGs in terms of predicted risk.

Secondary Objective

To build a novel predictive model solely on smartwatch ECG to predict risk for cardiomyopathy.

DETAILED DESCRIPTION:
The proposed study is looking to compare the 30 second ECG read from a smartwatch to the clinical ECG during a SJLIFE scheduled ECG appointment.

ELIGIBILITY:
Inclusion Criteria:

* SJLIFE participant and 22 years of age or older at time of enrollment
* Participant or legal guardian is able and willing to give informed consent
* At least 5 years after childhood cancer diagnosis

Exclusion Criteria:

* Been diagnosed with cardiomyopathy on previous SJLIFE ECG
* Currently on heart medication

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 1303 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Standard 12-lead ECG | Baseline
  To be obtained during SLIFE Human Performance Lab appointment. Participant will receive a resting (supine) 12-lead ECG using a GE Mac 2000 Resting ECG System (General Electric Healthcare, Milwaukee, WI, USA). This will be assessed with the Apple Smartwatch ECG recording to determine concordance of the two ECGs.
Apple Smartwatch ECG 30-second recording | Baseline
  To be obtained during the SLIFE Human Performance Lab appointment, collected immediately after recording of the standard 12-lead ECG. A study team member will place an Apple Smartwatch Series 7 on the participant's wrist. The participant will be instructed to start the ECG, which will be a 30-second recording process. Once captured, the data will be automatically transferred to the IOS application on the study iPhone. This will be assessed with the standard 12-lead ECG recording to determine concordance of the two ECGs.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Hudson, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols